CLINICAL TRIAL: NCT05666479
Title: Clinical Effectiveness of Continuous Blood Glucose Monitoring In Patients With Type 2 Diabetes Undergoing Orthopaedic Hip or Knee Replacement Surgery
Brief Title: CGM Monitoring in T2DM Patients Undergoing Orthopaedic Replacement Surgery
Status: Active, not recruiting | Type: Observational
Sponsor: Stony Brook University (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Igor Kravets, Associate Professor of Medicine, Stony Brook University
Other Study IDs: IRB2021-00351
Record Dates: First submitted 2022-12-17; First posted 2022-12-27 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Diabetes Mellitus, Type 2; Arthroplasty, Replacement, Hip; Arthroplasty, Replacement, Knee
Keywords: Type 2 Diabetes; Orthopaedic Hip Replacement; Orthopaedic Knee Replacement; Continuous Blood Glucose Monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Patients with Type 2 Diabetes Undergoing Orthopaedic Hip or Knee Replacement Surgery
  Interventions: Device: Dexcom G6 Pro Continuous Glucose Monitor (CGM)

INTERVENTIONS:
Device: Dexcom G6 Pro Continuous Glucose Monitor (CGM) — A DexCom G6 CGM will be implanted on the subject's abdomen contralateral to the surgical site (i.e. left abdomen for right knee or right hip replacements) no less than 30 cm from the surgical site. This CGM shall be termed "primary" for study purposes. Subjects will wear the primary DexCom G6 CGM for the entirety of the following 10-day timeline: 3/4-days pre-operative, day of hip or knee replacement surgery, and 5/6-day postoperative recovery.
  A second CGM will be implanted in subjects postoperatively while in the Post Anesthesia Care Unit (PACU). This CGM, termed "secondary" for study purposes, will be implanted immediately adjacent to the primary CGM. Subjects will wear the secondary DexCom CGM for the 7 days: day of hip or knee replacement surgery (postoperatively) and 5/6-day postoperative recovery.

SUMMARY:
The purpose of this study is to analyze the efficacy and accuracy of real-time continuous glucose monitoring devices (rtCGM) in patients with Type 2 diabetes undergoing inpatient elective hip or knee surgery in the pre-, peri-, and post-operative setting at Stony Brook University Hospital (SBUH).

ELIGIBILITY:
Inclusion Criteria:

* Greater than or equal to 18 years of age
* Scheduled for elective inpatient hip or knee replacement surgery at Stony Brook University Hospital (SBUH)
* Clinically diagnosed Type 2 Diabetes at least 6 months prior to surgery
* Literate and able to provide written informed consent
* Negative pregnancy test by serum or urine HCG at screening [as documented in subject's medical record) for women of childbearing potential (WCBP)]

Exclusion Criteria:

* Less than 18 years of age
* Not scheduled for elective inpatient hip or knee replacement surgery at SBUH
* No clinical diagnosis of Type 2 diabetes at least 6 months prior to surgery
* Not literate or unable to provide written informed consent
* Documented diagnosis of organ failure
* Documented diagnosis of chronic infection
* Documented diagnosis of any active malignancy
* Documented diagnosis of hepatic (liver) dysfunction or cirrhosis
* Pregnant by serum or urine HCG at screening [as documented in subject's medical record) for women of childbearing potential (WCBP)]

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with type 2 diabetes undergoing orthopaedic hip or knee replacement surgery.
Sampling Method: Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2022-09-09 (Actual); Primary Completion 2024-04-30 (Estimated); Study Completion 2024-09 (Estimated)

PRIMARY OUTCOMES:
Accuracy of Real-Time Continuous Glucose Monitoring | 10 days
  Analyze data from real-time continuous glucose monitoring and point-of-care glucose monitoring (POC-BG). rtCGM data will be matched and compared to POC-BG collected for standard clinical care in the pre-op and post-op settings (i.e. mealtimes, bedtime, and every 6 hours).

SECONDARY OUTCOMES:
Interference of Intraoperative Electrocautery on Real-Time Continuous Glucose Monitoring | 60-90 minutes
  Analyze intraoperative rtCGM. Electrocautery, a common surgical technique using electrical current to mitigate bleeding by thermal damage of tissue, may emit electrical pulses which adversely interfere with the measurement and/or data transmission of the rtCGM device. All data points collected during the 60-90-minute operative window will be analyzed for interference, aberrant, or missing values.
Assess Irreversible Damage/Interference of Real-Time Continuous Glucose Monitoring Devices Caused by Electrocautery | 6-7 days
  Assess irreversible damage/interference of rtCGMs caused by electrocautery. In the postoperative setting, a second rtCGM will be implanted on patients. Data sets between the two rtCGMs will be analyzed for statistically significant mean absolute relative difference (MARD).

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No